CLINICAL TRIAL: NCT02000817
Title: A Single Blind, Randomised, Placebo Controlled, Repeat Dose, Dose Escalating Study Investigating Safety, Tolerability Pharmacokinetics, Pharmacodynamics and the Beta-Cell Preserving Effect of Otelixizumab in New-Onset, Autoimmune Type 1 Diabetes Mellitus Patients
Brief Title: Investigation of Otelixizumab in New-Onset, Autoimmune Type 1 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 116505; 2013-003296-34 (EudraCT Number)
Record Dates: First submitted 2013-11-07; First posted 2013-12-04 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Beta Cell; Monoclonal Antibody; Otelixizumab; Cytokine Release Syndrome; Epstein-Barr Virus; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Cytokine Release Syndrome; Epstein-Barr Virus Infections; Diabetes Mellitus | interventions — otelixizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Otelixizumab 9 mg (Experimental): Each subject will receive otelixizumab 1.5 mg diluted with 0.9% weight /volume sodium chloride intravenously daily for 6 consecutive days (cumulative dose-9 mg)
  Interventions: Biological: Otelixizumab
- Otelixizumab 18 mg (Experimental): Each subject will receive otelixizumab 3 mg diluted with 0.9% weight /volume sodium chloride intravenously daily for 6 consecutive days (cumulative dose-18 mg)
  Interventions: Biological: Otelixizumab
- Otelixizumab 27 mg (Experimental): Each subject will receive otelixizumab 4.5 mg diluted with 0.9% weight /volume sodium chloride intravenously daily for 6 consecutive days (cumulative dose-27 mg)
  Interventions: Biological: Otelixizumab
- Otelixizumab 36 mg (Experimental): Each subject will receive otelixizumab 1.5 mg diluted with 0.9% weight /volume sodium chloride intravenously daily for 6 consecutive days (cumulative dose-36 mg)
  Interventions: Biological: Otelixizumab
- Placebo (Placebo Comparator): Each subject will receive otelixizumab matching placebo diluted with 0.9% weight /volume sodium chloride intravenously daily for 6 consecutive days
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Otelixizumab — Otelixizumab is available at unit dose strength of 5 milligram/mL provided as 1 mL solution per vial to be diluted to 0.1 mg/mL in 0.9% sodium chloride. The 0.1 mg/mL solution is to be administered by intravenous infusion using a syringe pump and an in-line 0.2 micron filter by study personnel following specified regimens
  Arms: Otelixizumab 18 mg; Otelixizumab 27 mg; Otelixizumab 36 mg; Otelixizumab 9 mg
Biological: Placebo — Placebo is available 0.9% w/v sodium chloride
  Arms: Placebo

SUMMARY:
The aim of this Phase I/IIa study is to identify a safe and tolerable dosage regimen of intravenously administered otelixizumab. In addition, the C-peptide decline in new onset type 1 diabetes mellitus (NOT1DM) patients and possible immunological mechanisms will be investigated with a view to identifying trends and early immunological biomarkers which could predict response in halting/slowing Beta-cell destruction in this patient population.

This exploratory study will explore the safety and tolerability between the well tolerated but non-efficacious cumulative dose of 3.1 mg and a cumulative dose of 48 mg at which efficacy based on C-peptide analysis was demonstrated, albeit with evidence of Epstein Barr Virus (EBV) reactivation and Cytokine Release Syndrome (CRS). Exploration of the tolerability dose response is considered a necessary first step to determining the therapeutic index of otelixizumab.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 16 and 27 years of age inclusive, at the time of signing the informed consent.

NOTE: Subjects aged 16 to 17 years must be Tanner Stage >= 2. All subjects must weigh at least 31 kg.

* Diagnosis of diabetes mellitus (DM) according to Amerrican Diabetes Association (ADA) and World Health Organization (WHO) criteria and consistent with Type 1a (autoimmune) Diabetes Mellitus (T1DM), with an interval of approximately 28 days (not more than 32 days) between the initial diagnosis and the first dose of study drug). Written documentation of the diagnosis of DM, including the date of diagnosis, must be obtained from the diagnosing physician.
* Currently requires insulin treatment for T1DM and has received intensive insulin therapy for at least 7 days prior to screening.
* Positive for at least one auto-antibody associated with T1DM: antibody to glutamic acid decarboxylase (anti GAD), antibody to protein tyrosine phosphatase-like protein (anti IA 2), antibody to islet-cell antigen (ICA) or ZnT8 Autoantibody.
* Evidence of residual functioning Beta-cells as measured by mixed meal stimulated C peptide peak level >= 0.2 nanomole/litre (nmol/L).
* A female subject is eligible to participate if she has a negative pregnancy test as determined by a urine hCG test at screening or prior to dosing and agrees to use one of the contraception methods listed in study protocol. Female subjects must agree to use contraception for 2 weeks prior to dosing and for 60 days after the last dose of study drug or has only same-sex partners (refrains from heterosexual intercourse), when this is her preferred and usual lifestyle.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in study protocol. This criterion must be followed from 2 weeks prior to dosing and for 60 days after the last dose of study drug.
* Willing to follow the procedures outlined in the protocol.
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2xupper limit of normal (ULN); alkaline phosphatase and bilirubin <= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Subjects eligible for enrolment in the study must meet all of the following criteria: QTc <450msec or QTc <480msec for patients with bundle branch block. The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF), or another method, machine or manual overread. For subject eligibility and withdrawal, QTcF will be used. For purposes of data analysis, QTcF will be used as primary. The QTc should be based on single or averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period.
* Screening total lymphocyte counts within the normal range in two separate samples taken at least three days apart (eg screening and Day -1).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form. In the case of minors (under 18 years) written informed consent must also be obtained from a parent or Legally Acceptable Representative (LAR).

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or core antibody or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive test for Human Immunodeficiency Virus (HIV) 1 and/or 2 antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new investigational drugs within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within a 3 month period.
* Lactating females.
* Subject is mentally or legally incapacitated.
* History of thrombocytopenia.
* The subject has received immunizationion with a vaccine within 4 weeks before the first dose of study drug or requires a vaccine within 30 days after the last dose of study drug
* The subject has had significant systemic infection during the 6 weeks before the first dose of study drug (e.g., infection requiring hospitalization, major surgery, or intravenous (i.v.) antibiotics to resolve; other infections, e.g., bronchitis, sinusitis, localized cellulitis, candidiasis, or urinary tract infections, must be assessed on a case-by-case basis by the investigator regarding whether they are serious enough to warrant exclusion).
* Current or prior malignancy, other than non-melanoma skin cancer.
* Patient has undergone a splenectomy
* Radiological evidence of active tuberculosis (TB).
* Significant and/or active disease in any body system likely to increase the risk to the subject or interfere with the subject's participation in or completion of the study. Examples of significant diseases include, but are not limited to, coronary artery disease, congestive heart failure, uncontrolled hypertension, renal failure, emphysema, history of bleeding peptic ulcers, history of seizure(s), addiction to illicit drugs, and alcohol abuse.
* Clinically significant (based on Investigator's discretion in consultation with the Medical Monitor if second opinion required) abnormal laboratory values during the Screening period, other than those due to T1DM. A clinically significant abnormal value will not result in exclusion if, upon re test, the abnormality is resolved or becomes clinically insignificant.
* Positive EBV capsid Ab IgM in absence of a positive EBV EBNA Ab IgG
* EBV viral load of> 10,000 copies per 10^6 peripheral blood mononuclear cells (PBMCs) as determined by quantitative polymerase chain reaction (qPCR)
* Immunoglobulin G (IgG) negative for EBV.
* A positive result on an Immuno-Assay test for syphilis; and, if result of Immuno-assay test is positive, then a confirmatory test will be performed.
* Have used any atypical antipsychotic drug (e.g., risperidone, quetiapine, or clozapine) within the 30 days before signing the Informed Consent Form (ICF).
* Have previously received otelixizumab or any other anti cluster of differentiation (CD)3 monoclonal antibody, e.g. muromonab, or teplizumab, and are not willing to refrain from using any such antibody for the planned duration of study participation (2 years after the last dose of study drug).
* Previous or current exposure to biologic cell-depleting therapies (e.g. anti-CD11a, anti-CD22, anti-CD20, anti- B lymphocyte stimulator/ B-cell activating factor (BLyS/BAFF), anti-CD3, anti-CD5, anti-CD52) including investigational agents, and planning to use any such antibody for the planned duration of study participation (2 years after the last dose of study drug).
* Predisposition to thromboembolic disease, or thromboembolic event (excluding superficial) in the past 12 months.
* Is currently receiving corticoid treatment or has received systemic corticoid treatment within a month of screening,
* History of Graves disease
* Prior allergic reaction, including anaphylaxis, to any human, humanised, chimeric, or rodent antibody.
* Have undergone any major surgical procedure within 30 days before the first dose of study drug, and/or planning to undergo any such surgery within 3 months after the last dose of study drug.
* Any condition or situation that, in the investigator's judgment, is likely to cause the subject to be unable or unwilling to participate in study procedures or to complete all scheduled assessments.

Ages: 16 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Belgium (5):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège

REFERENCES:
- [Derived] Keymeulen B, van Maurik A, Inman D, Oliveira J, McLaughlin R, Gittelman RM, Roep BO, Gillard P, Hilbrands R, Gorus F, Mathieu C, Van de Velde U, Wisniacki N, Napolitano A. A randomised, single-blind, placebo-controlled, dose-finding safety and tolerability study of the anti-CD3 monoclonal antibody otelixizumab in new-onset type 1 diabetes. Diabetologia. 2021 Feb;64(2):313-324. doi: 10.1007/s00125-020-05317-y. Epub 2020 Nov 4. PMID 33145642
- [Derived] Vlasakakis G, Napolitano A, Barnard R, Brown K, Bullman J, Inman D, Keymeulen B, Lanham D, Leirens Q, MacDonald A, Mezzalana E, Page K, Patel M, Savage CO, Zamuner S, van Maurik A. Target engagement and cellular fate of otelixizumab: a repeat dose escalation study of an anti-CD3epsilon mAb in new-onset type 1 diabetes mellitus patients. Br J Clin Pharmacol. 2019 Apr;85(4):704-714. doi: 10.1111/bcp.13842. Epub 2019 Feb 5. PMID 30566758

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a multi-centered, single-blind, randomized, placebo-controlled 6 Day repeat dose study to investigate the safety, tolerability, pharmacokinetics, pharmacodynamics, efficacy and immunological profile of intravenously administered Otelixizumab (OTX) in New Onset Type 1 Diabetes Mellitus participants.
Pre-assignment Details: A total of 30 participants were enrolled at different centers in Belgium, which was conducted from 12-Mar-2014 to 27-Sep-2018.
Groups:
- Placebo: Participants received 0.9% weight/volume Sodium Chloride solution for injection daily for 6 Days
- Otelixizumab 9 mg: Participants received 1.5 mg of OTX (intravenous solution for infusion) daily for 6 Days
- Otelixizumab 18 mg: Participants received 3 mg of OTX (intravenous solution for infusion) daily for 6 Days
- Otelixizumab 27 mg: Participants received 4.5 mg of OTX (intravenous solution for infusion) daily for 6 Days
Period: Overall Study
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Started | 6 | 9 | 8 | 7
Completed | 4 | 8 | 7 | 7
Not Completed | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population comprised of participants who received at least one dose of study treatment. 1 participant withdrew after being randomized, prior to receiving any treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg | Total
Number analyzed (Participants) | 5 | 9 | 8 | 7 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] — Safety Population comprised of participants who received at least one dose of study treatment. 1 participant withdrew after being randomized, prior to receiving any treatment.
  Years | 24.8 (4.44) | 22.4 (2.13) | 20.5 (4.31) | 22.1 (3.98) | 22.2 (3.77)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population comprised of participants who received at least one dose of study treatment. 1 participant withdrew after being randomized, prior to receiving any treatment.
  Participants
    Female | 2 | 3 | 3 | 2 | 10
    Male | 3 | 6 | 5 | 5 | 19
Race/Ethnicity, Customized [Number; unit: Count of Participants] — Safety Population comprised of participants who received at least one dose of study treatment. 1 participant withdrew after being randomized, prior to receiving any treatment.
  Count of Participants
    WHITE | 5 | 9 | 8 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) Related to Cytokine Release Syndrome (CRS)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. On treatment AEs have been reported. Safety Population comprised of all participants who received at least one dose of study treatment.
Time Frame: Up to Day 14
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Participants | 5 | 9 | 8 | 7

2. Primary Outcome: Epstein-Barr Virus (EBV) Viral Load Detection
Description: Blood samples were collected for analysis of EBV viral load and detection was done by polymerase chain reaction (PCR).
Time Frame: Week 3, Week 6, Week 8, Week 12, Week 24 and Week 96
Population: Safety population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies per million cells
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Copies per million cells
  Week 3, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Week 3, n=5, 8, 8, 7 | 12.0 (32806.06) | 438.5 (193067.66) | 4266.1 (306867.44) | 64870.6 (723.66)
  Week 6, n=4, 9, 8, 7: number analyzed (Participants) | 4 | 9 | 8 | 7
  Week 6, n=4, 9, 8, 7 | 28.1 (178623.77) | 20.5 (77662.74) | 398.2 (131086.12) | 974.2 (19777.11)
  Week 8, n=5, 9, 7, 5: number analyzed (Participants) | 5 | 9 | 7 | 5
  Week 8, n=5, 9, 7, 5 | 3.5 (4755.63) | 8.9 (22969.48) | 17.0 (55312.01) | 24.3 (3060948.75)
  Week 12, n=4, 9, 8, 6: number analyzed (Participants) | 4 | 9 | 8 | 6
  Week 12, n=4, 9, 8, 6 | 4.7 (12491.55) | 15.8 (21359.16) | 5.5 (15292.04) | 33.2 (227953.09)
  Week 24, n=4, 9, 7, 7: number analyzed (Participants) | 4 | 9 | 7 | 7
  Week 24, n=4, 9, 7, 7 | 1.0 (0.00) | 39.3 (52129.25) | 15.9 (39905.91) | 2.9 (4732.52)
  Week 96, n=4, 9, 7, 7: number analyzed (Participants) | 4 | 9 | 7 | 7
  Week 96, n=4, 9, 7, 7 | 1.0 (0.00) | 2.3 (2166.53) | 3.3 (13653.67) | 5.9 (9925.87)

3. Primary Outcome: Number of Participants With Abnormal Laboratory Results
Description: Blood samples were collected to analyze the laboratory parameters which included alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), bilirubin, calcium, chloride, creatinine, direct bilirubin, glucose, potassium, protein, sodium, urate, urea nitrogen, basophil, eosinophil, mean corpuscular haemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), mean corpuscular volume (MCV), erythrocytes, haematocrit, haemoglobin, leukocytes, lymphocytes, monocytes, neutrophils, platelets and reticulocytes.
Time Frame: Up to Month 24
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Participants
  ALT, Low, n= 5, 9, 8, 7 | 0 | 0 | 0 | 1
  ALT, High, n= 5, 9, 8, 7 | 2 | 5 | 6 | 4
  Albumin, Low, n= 5, 9, 8, 7 | 4 | 5 | 2 | 3
  Albumin, High, n= 5, 9, 8, 7 | 1 | 4 | 1 | 0
  ALP, Low, n= 5, 9, 8, 7 | 3 | 0 | 1 | 1
  ALP, High, n= 5, 9, 8, 7 | 0 | 1 | 0 | 1
  AST, Low, n= 5, 9, 8, 7 | 1 | 0 | 1 | 0
  AST, High, n= 5, 9, 8, 7 | 1 | 4 | 5 | 5
  Bilirubin, Low, n= 5, 9, 8, 7 | 2 | 2 | 2 | 1
  Bilirubin, High, n= 5, 9, 8, 7 | 0 | 1 | 2 | 2
  Calcium, Low, n= 5, 9, 8, 7 | 1 | 5 | 5 | 1
  Calcium, High, n= 5, 9, 8, 7 | 0 | 1 | 1 | 0
  Chloride, Low, n= 5, 9, 8, 7 | 0 | 2 | 0 | 1
  Chloride, High, n= 5, 9, 8, 7 | 3 | 5 | 5 | 3
  Creatinine, Low, n= 5, 9, 8, 7 | 1 | 0 | 2 | 1
  Creatinine, High, n= 5, 9, 8, 7 | 0 | 3 | 0 | 0
  Direct Bilirubin, Low, n= 1, 5, 4, 5: number analyzed (Participants) | 1 | 5 | 4 | 5
  Direct Bilirubin, Low, n= 1, 5, 4, 5 | 0 | 0 | 0 | 0
  Direct Bilirubin, High, n= 1, 5, 4, 5: number analyzed (Participants) | 1 | 5 | 4 | 5
  Direct Bilirubin, High, n= 1, 5, 4, 5 | 0 | 0 | 0 | 1
  Glucose, Low, n= 5, 9, 8, 7 | 4 | 0 | 0 | 2
  Glucose, High, n= 5, 9, 8, 7 | 2 | 2 | 1 | 3
  Potassium, Low, n= 5, 9, 8, 7 | 0 | 3 | 3 | 2
  Potassium, High, n= 5, 9, 8, 7 | 0 | 0 | 1 | 0
  Protein, Low, n= 5, 9, 8, 7 | 2 | 3 | 7 | 3
  Protein, High, n= 5, 9, 8, 7 | 0 | 0 | 0 | 0
  Sodium, Low, n= 5, 9, 8, 7 | 1 | 0 | 1 | 2
  Sodium, High, n= 5, 9, 8, 7 | 0 | 3 | 1 | 0
  Urate, Low, n= 5, 9, 8, 7 | 1 | 6 | 1 | 6
  Urate, High, n= 5, 9, 8, 7 | 0 | 0 | 0 | 1
  Urea Nitrogen, Low, n= 5, 9, 8, 7 | 2 | 5 | 3 | 2
  Urea Nitrogen, High, n= 5, 9, 8, 7 | 1 | 2 | 2 | 1
  Basophils, Low, n= 5, 9, 8, 7 | 0 | 1 | 0 | 0
  Basophils, High, n= 5, 9, 8, 7 | 0 | 0 | 1 | 0
  Eosinophils, Low, n= 5, 9, 8, 7 | 0 | 1 | 0 | 0
  Eosinophils, High, n= 5, 9, 8, 7 | 3 | 2 | 2 | 1
  MCHC, Low, n= 5, 9, 8, 7 | 2 | 1 | 2 | 2
  MCHC, High, n= 5, 9, 8, 7 | 1 | 5 | 4 | 4
  MCH, Low, n= 5, 9, 8, 7 | 0 | 2 | 4 | 3
  MCH, High, n= 5, 9, 8, 7 | 0 | 0 | 1 | 0
  MCV, Low, n= 5, 9, 8, 7 | 0 | 3 | 3 | 2
  MCV, High, n= 5, 9, 8, 7 | 0 | 0 | 0 | 0
  Erythrocytes, Low, n= 5, 9, 8, 7 | 4 | 6 | 6 | 4
  Erythrocytes, High, n= 5, 9, 8, 7 | 0 | 2 | 1 | 0
  Hematocrit, Low, n= 5, 9, 8, 7 | 4 | 5 | 7 | 2
  Hematocrit, High, n= 5, 9, 8, 7 | 1 | 0 | 0 | 0
  Hemoglobin, Low, n= 5, 9, 8, 7 | 5 | 6 | 5 | 4
  Hemoglobin, High, n= 5, 9, 8, 7 | 0 | 2 | 0 | 0
  Leukocytes, Low, n= 5, 9, 8, 7 | 0 | 5 | 2 | 2
  Leukocytes, High, n= 5, 9, 8, 7 | 3 | 1 | 1 | 1
  Lymphocytes, Low, n= 5, 9, 8, 7 | 0 | 9 | 7 | 7
  Lymphocytes, High, n= 5, 9, 8, 7 | 1 | 1 | 2 | 3
  Monocytes, Low, n= 5, 9, 8, 7 | 0 | 1 | 0 | 2
  Monocytes, High, n= 5, 9, 8, 7 | 0 | 0 | 0 | 1
  Neutrophils, Low, n= 5, 9, 8, 7 | 0 | 2 | 2 | 2
  Neutrophils, High, n= 5, 9, 8, 7 | 2 | 1 | 2 | 2
  Platelets, Low, n= 5, 9, 8, 7 | 0 | 2 | 3 | 2
  Platelets, High, n= 5, 9, 8, 7 | 0 | 0 | 2 | 0
  Reticulocytes, Low, n= 1, 3, 4, 4: number analyzed (Participants) | 1 | 3 | 4 | 4
  Reticulocytes, Low, n= 1, 3, 4, 4 | 0 | 1 | 0 | 0
  Reticulocytes, High, n= 1, 3, 4, 4: number analyzed (Participants) | 1 | 3 | 4 | 4
  Reticulocytes, High, n= 1, 3, 4, 4 | 0 | 2 | 1 | 1

4. Primary Outcome: Number of Participants With Increase in QT Interval Corrected for Heart Rate (QTc)
Description: 12-lead electrocardiograms (ECGs) were obtained in semi-supine position after 5 minutes rest for the participants at indicated time points to measure QTc.
Time Frame: Up to Month 24
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Participants
  QTc Interval (Bazett's), Increase >60 millisec | 0 | 0 | 0 | 0
  QTc Interval (Fridericia), Increase >60 millisec | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Vital Sign Results
Description: Vital signs were measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Vital signs included systolic, diastolic blood pressure, pulse rate and respiratory rate
Time Frame: Up to Month 24
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Participants
  Systolic Blood Pressure, Low | 1 | 1 | 2 | 1
  Systolic Blood Pressure, High | 1 | 0 | 1 | 1
  Diastolic Blood Pressure, Low | 2 | 5 | 4 | 1
  Diastolic Blood Pressure, High | 0 | 0 | 1 | 0
  Pulse Rate, Low | 0 | 0 | 0 | 1
  Pulse Rate, High | 1 | 2 | 3 | 2
  Respiratory Rate, Low | 0 | 1 | 0 | 0
  Respiratory Rate, High | 0 | 0 | 0 | 0

6. Secondary Outcome: Free Serum Otelixizumab Concentrations by Treatment
Description: Blood samples were collected at designated timepoints. Free serum Otelixizumab concentrations were calculated by linear and semi-logarithmic individual serum concentration-time profiles. Fully treated population comprised of all randomized participants who received the full 6 days of treatment based on actual exposure data. NA indicates that data could not be calculated as >30% of samples were below the limit of quantification.
Time Frame: Pre-dose on Day 1,2,3,4,5,6 and 14; 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 9 hours, 16 hours post-dose on Day 1, and 1 hour post-dose on Day 6.
Population: Fully Treated population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 8 | 8 | 6
Nanogram per milliliter (ng/mL)
  Day 1, Pre-dose, n=8, 8, 6 | 0.000 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 0.000 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 0.000 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification.
  Day 1, 30 minutes, n=8, 8, 6 | 0.000 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 0.444 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 7.387 (4.8946)
  Day 1, 1 hour, n=8, 8, 6 | 0.513 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 2.963 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 12.542 (7.9086)
  Day 1, 2 hours, n=8, 8, 6 | 2.995 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 7.606 (6.1836) | 23.598 (14.4526)
  Day 1, 4 hours, n=7, 8, 6: number analyzed (Participants) | 7 | 8 | 6
  Day 1, 4 hours, n=7, 8, 6 | 6.600 (5.2773) | 15.929 (9.8903) | 41.457 (26.3827)
  Day 1, 6 hours, n=8, 8, 6 | 11.870 (5.0544) | 24.899 (14.5630) | 100.148 (79.4845)
  Day 1, 8 hours, n=8, 7, 6: number analyzed (Participants) | 8 | 7 | 6
  Day 1, 8 hours, n=8, 7, 6 | 70.088 (153.2593) | 37.657 (19.8741) | 146.298 (95.4089)
  Day 1, 9 hours, n=7, 8, 6: number analyzed (Participants) | 7 | 8 | 6
  Day 1, 9 hours, n=7, 8, 6 | 18.494 (6.0716) | 102.865 (111.2186) | 402.173 (246.4271)
  Day 1, 16 hours, n=7, 8, 6: number analyzed (Participants) | 7 | 8 | 6
  Day 1, 16 hours, n=7, 8, 6 | 0.000 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 30.758 (23.3494) | 212.487 (144.0899)
  Day 2, Pre-Dose, n=8, 8, 6 | 0.000 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 7.329 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 112.020 (124.1743)
  Day 3, Pre-Dose, n=8, 8, 6 | 0.000 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 36.051 (35.6464) | 420.228 (344.7569)
  Day 4, Pre-Dose, n=8, 8, 6 | 0.523 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 114.993 (152.7864) | 829.148 (473.9342)
  Day 5, Pre-Dose, n=8, 8, 6 | 9.550 (16.2697) | 213.305 (257.3174) | 1088.808 (542.8032)
  Day 6, Pre-Dose, n=8, 8, 6 | 4.416 (3.2896) | 174.448 (258.4873) | 1386.008 (623.1118)
  Day 6, 1 hour, n=8, 8, 6 | 413.488 (262.5248) | 2048.336 (1889.7194) | 2868.735 (771.5457)
  Day 14, n=7, 8, 5: number analyzed (Participants) | 7 | 8 | 5
  Day 14, n=7, 8, 5 | 0.523 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 0.899 (NA) — NA indicates that data could not be calculated as it was below the limit of quantification. | 12.474 (8.7977)

7. Secondary Outcome: Change From Baseline in C-Peptide Weighted Mean (Area Under Curve From 0 to 120 Minutes [AUC0-120 Minutes]) From Mixed Meal Tolerance Test
Description: Blood samples were collected at indicated time points to assess levels of C-peptide. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Mixed meal-stimulated C-peptide AUC was calculated from area under C-peptide/time curve from time 0 to 120 minutes, using trapezoidal rule. ITT treated population comprised of all randomized participants who received at least one dose of study treatment.
Time Frame: Baseline (Day-1), Month 3, Month 6, Month 12, Month 18 and Month 24
Population: Intent-To-Treat (ITT) treated population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanomoles minute per liter
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Nanomoles minute per liter
  Month 3, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Month 3, n=5, 8, 8, 7 | 0.175 (0.0797) | 0.255 (0.2852) | 0.118 (0.2462) | 0.153 (0.1312)
  Month 6, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Month 6, n=5, 8, 8, 7 | 0.118 (0.0895) | 0.147 (0.3215) | -0.185 (0.2148) | 0.076 (0.2788)
  Month 12, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Month 12, n=5, 8, 8, 7 | -0.103 (0.0552) | 0.023 (0.3145) | -0.215 (0.2597) | -0.016 (0.3689)
  Month 18, n=5, 8, 7, 7: number analyzed (Participants) | 5 | 8 | 7 | 7
  Month 18, n=5, 8, 7, 7 | -0.278 (0.1142) | 0.015 (0.3903) | -0.295 (0.3105) | -0.201 (0.3132)
  Month 24, n=4, 7, 7, 7: number analyzed (Participants) | 4 | 7 | 7 | 7
  Month 24, n=4, 7, 7, 7 | -0.296 (0.0962) | -0.042 (0.2905) | -0.349 (0.3917) | -0.165 (0.3729)

8. Secondary Outcome: Change From Baseline in Glucose Weighted Mean (Area Under Curve From 0 to 120 Minutes, AUC0-120 Minutes) From Mixed Meal Tolerance Test
Description: Blood samples were collected at indicated time points to assess levels of glucose. Day -1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Mixed meal-stimulated glucose was calculated from area under the glucose /time curve from time 0 to 120 minutes, using trapezoidal rule.
Time Frame: Baseline (Day-1), Month 3, Month 6, Month 12, Month 18 and Month 24
Population: ITT treated population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Millmoles minute per liter
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Millmoles minute per liter
  Month 3, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Month 3, n=5, 8, 8, 7 | 1.382 (1.5801) | -0.550 (1.7140) | 0.999 (3.3953) | 0.641 (3.0009)
  Month 6, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Month 6, n=5, 8, 8, 7 | 1.423 (2.9999) | -1.041 (1.5506) | 0.643 (4.1751) | 0.749 (2.7698)
  Month 12, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Month 12, n=5, 8, 8, 7 | 2.314 (2.2718) | 0.067 (2.0492) | 1.875 (2.7440) | 1.842 (3.2408)
  Month 18, n=5, 8, 7, 7: number analyzed (Participants) | 5 | 8 | 7 | 7
  Month 18, n=5, 8, 7, 7 | 3.142 (3.2172) | 1.159 (2.4073) | 2.676 (3.0803) | 3.942 (1.9745)
  Month 24, n=4, 7, 7, 7: number analyzed (Participants) | 4 | 7 | 7 | 7
  Month 24, n=4, 7, 7, 7 | 4.029 (1.2365) | -1.807 (2.1615) | 2.557 (3.9428) | 3.435 (2.3714)

9. Secondary Outcome: Change From Baseline in C-Peptide Weighted Mean (Area Under Curve From 60 to 140 Minutes, [AUC 60-140 Minutes]) From Hyperglycemic Clamp Test
Description: Blood samples were collected at indicated time points to assess levels of C-peptide during hyperglycemic (H) phase. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from specified time point value. C-peptide AUC was calculated from area under C-peptide/time curve from time H60 to H140 minutes.
Time Frame: Baseline (Day-1), Month 6, Month 24
Population: ITT treated population. Only those participants with data available at specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanomoles minute per liter
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Nanomoles minute per liter
  Month 6, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Month 6, n=5, 8, 8, 7 | -0.037 (0.2107) | 0.105 (0.2520) | -0.201 (0.2643) | 0.006 (0.3011)
  Month 24, n=4, 5, 7, 7: number analyzed (Participants) | 4 | 5 | 7 | 7
  Month 24, n=4, 5, 7, 7 | -0.423 (0.1630) | -0.273 (0.1552) | -0.373 (0.2308) | -0.344 (0.3397)

10. Secondary Outcome: Change From Baseline in Glucose Weighted Mean (Area Under Curve From 60 to 140 Minutes, AUC60-140 Minutes) From Hyperglycemic Clamp Test
Description: Blood samples were collected at indicated time points to assess levels of glucose during hyperglycemic (H) phase. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Glucose AUC was calculated from area under the C-peptide/time curve from time H60 to H140 minutes.
Time Frame: Baseline (Day-1), Month 6 and Month 24
Population: ITT treated population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Millmoles minute per liter
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Millmoles minute per liter
  Month 6, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Month 6, n=5, 8, 8, 7 | 0.645 (1.0094) | 0.415 (1.3255) | 0.723 (1.5955) | 1.074 (0.6264)
  Month 24, n=4, 5, 7, 7: number analyzed (Participants) | 4 | 5 | 7 | 7
  Month 24, n=4, 5, 7, 7 | 1.346 (1.1063) | -0.501 (3.2542) | 0.094 (2.2642) | 1.095 (1.3972)

11. Secondary Outcome: Change From Baseline in Insulin Sensitivity (IS) Index From Hyperglycemic Clamp Test
Description: Insulin sensitivity index is defined as the ratio of glucose metabolized and average insulin concentration multiplied by 100 by hyperglycemic clamp test. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day-1), Month 6, Month 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: (100*mmol*l)/(pmol*kg*min)
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
(100*mmol*l)/(pmol*kg*min)
  Month 6, n=5, 8, 7, 6: number analyzed (Participants) | 5 | 8 | 7 | 6
  Month 6, n=5, 8, 7, 6 | -0.0003 (0.00130) | -0.0000 (0.00030) | -0.0002 (0.00197) | -0.0002 (0.00066)
  Month 24, n=4, 4, 6, 6: number analyzed (Participants) | 4 | 4 | 6 | 6
  Month 24, n=4, 4, 6, 6 | 0.0037 (0.00591) | -0.0006 (0.00344) | -0.0013 (0.01299) | 0.0023 (0.00351)

12. Secondary Outcome: Change From Baseline in Mean Daily Insulin Use
Description: Participants were asked to record their daily insulin usage thoroughly and accurately in a diary from 7 days prior to study visit. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day-1), Week 2, Week 3, Week 6, Week 8, Week 12, Week 24, Week 36, Week 48, Week 72 and Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: International unit
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
International unit
  Week 2, n=5, 8, 7, 6: number analyzed (Participants) | 5 | 8 | 7 | 6
  Week 2, n=5, 8, 7, 6 | -0.0901 (0.05997) | -0.0265 (0.07580) | 0.0941 (0.12919) | -0.0741 (0.08855)
  Week 3, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Week 3, n=5, 8, 8, 7 | -0.1504 (0.06424) | -0.0424 (0.08708) | 0.0706 (0.14989) | -0.0440 (0.08753)
  Week 6, n=5, 4, 8, 7: number analyzed (Participants) | 5 | 4 | 8 | 7
  Week 6, n=5, 4, 8, 7 | -0.1727 (0.05431) | -0.1009 (0.12893) | -0.0332 (0.19098) | -0.1090 (0.11777)
  Week 8, n=4, 7, 5, 6: number analyzed (Participants) | 4 | 7 | 5 | 6
  Week 8, n=4, 7, 5, 6 | -0.1566 (0.07033) | -0.1514 (0.15364) | -0.0666 (0.21066) | -0.1492 (0.14713)
  Week 12, n=4, 8, 8, 7: number analyzed (Participants) | 4 | 8 | 8 | 7
  Week 12, n=4, 8, 8, 7 | -0.1850 (0.08007) | -0.1629 (0.14706) | -0.1115 (0.16950) | -0.1850 (0.20173)
  Week 24, n=5, 8, 5, 7: number analyzed (Participants) | 5 | 8 | 5 | 7
  Week 24, n=5, 8, 5, 7 | -0.1449 (0.09069) | -0.1168 (0.20181) | 0.0298 (0.13942) | -0.1678 (0.17308)
  Week 36, n=4, 8, 7, 7: number analyzed (Participants) | 4 | 8 | 7 | 7
  Week 36, n=4, 8, 7, 7 | -0.0776 (0.13492) | -0.0673 (0.26527) | 0.0701 (0.20840) | -0.1114 (0.21943)
  Week 48, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Week 48, n=5, 8, 8, 7 | -0.1221 (0.16778) | -0.0936 (0.24246) | 0.0970 (0.15473) | -0.1155 (0.25461)
  Week 72, n=5, 8, 7, 5: number analyzed (Participants) | 5 | 8 | 7 | 5
  Week 72, n=5, 8, 7, 5 | -0.1000 (0.23378) | 0.0172 (0.43320) | 0.1088 (0.07406) | 0.0807 (0.27375)
  Week 96, n=4, 6, 7, 7: number analyzed (Participants) | 4 | 6 | 7 | 7
  Week 96, n=4, 6, 7, 7 | -0.0390 (0.34885) | -0.0811 (0.34104) | 0.1131 (0.16596) | 0.1117 (0.19080)

13. Secondary Outcome: Change From Baseline in Hemoglobin A1c
Description: Hemoglobin A1C levels were measured at indicated time points. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day-1), Month 6, Month 12 and Month 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Percentage of HbA1c
  Month 6, n=5, 8, 8, 7: number analyzed (Participants) | 5 | 8 | 8 | 7
  Month 6, n=5, 8, 8, 7 | -3.26 (1.119) | -2.29 (1.883) | -0.68 (2.437) | -2.04 (2.141)
  Month 12, n=5, 9, 8, 7 | -3.26 (1.665) | -2.10 (2.125) | -1.15 (1.384) | -1.60 (2.985)
  Month 24, n=4, 9, 7, 7: number analyzed (Participants) | 4 | 9 | 7 | 7
  Month 24, n=4, 9, 7, 7 | -2.53 (2.445) | -2.23 (1.736) | -0.33 (2.075) | -1.41 (2.174)

14. Secondary Outcome: Absolute Body Weight
Description: Body weight was measured at indicated time points.
Time Frame: Day-1, Month 12, Month 18 and Month 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Kilogram
  Day -1, n=5, 9, 8, 7 | 65.22 (10.608) | 72.84 (16.118) | 64.19 (9.545) | 65.27 (8.714)
  Month 12, n=5, 9, 8, 7 | 70.24 (12.691) | 75.86 (15.503) | 64.58 (9.851) | 67.96 (8.373)
  Month 18, n=5, 9, 7, 7: number analyzed (Participants) | 5 | 9 | 7 | 7
  Month 18, n=5, 9, 7, 7 | 70.44 (13.209) | 75.22 (16.504) | 63.56 (8.658) | 68.97 (10.167)
  Month 24, n=4, 9, 7, 7: number analyzed (Participants) | 4 | 9 | 7 | 7
  Month 24, n=4, 9, 7, 7 | 66.98 (11.226) | 75.82 (17.507) | 63.71 (8.037) | 69.79 (8.689)

15. Secondary Outcome: Time-normalized Number of Hypoglycemic and Hyperglycemic Events
Description: As per American Diabetes Association (ADA), hypoglycemia is defined as blood glucose level <= 70 milligram/deciliter (mg/dl) and hyperglycemia is defined as blood glucose level > 250 mg/dL. Hypoglycaemic and hyperglycaemic events will be recorded in a diary whenever they occur, along with the start and stop dates. Mean number of events is defined as the average number of events reported per subject. Normalization is expressed by dividing number of events by length of reporting period in month (1 month = 30 days).
Time Frame: Up to Month 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 4 | 9 | 7 | 7
Number of events
  Hypoglycemia | 14.13 (3.533) | 21.45 (2.383) | 7.74 (1.105) | 24.55 (3.508)
  Hyperglycemia | 2.79 (0.698) | 11.03 (1.225) | 14.13 (2.019) | 8.48 (1.211)

16. Secondary Outcome: Relative Change From Baseline in Percentage (%) in CD4+ Cells
Description: Whole blood samples were collected and analyzed by flow cytometry. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Relative change from Baseline (percentage) was calculated as change from Baseline relative to Baseline in percentage.
Time Frame: Day 1 (30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 9 hours, 12 hours, 16 hours), Day 2, Day 3, Day 4, Day 5, Day 6 (1 hour), Day 14
Population: Fully treated population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Percentage
  Day 1, 30 minutes, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 30 minutes, n=5, 7, 8, 6 | -2.2331 (8.06090) | 15.7568 (9.45733) | 22.3101 (11.38275) | 37.9286 (7.06740)
  Day 1, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 1 hour, n=5, 7, 8, 6 | -0.9229 (3.79426) | 24.8673 (8.97161) | 33.2356 (10.06318) | 40.8432 (17.12371)
  Day 1, 2 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 2 hours, n=5, 7, 8, 6 | 4.6329 (10.59418) | 32.0976 (13.50078) | 42.2579 (11.17916) | 54.2045 (9.65956)
  Day 1, 4 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 4 hours, n=5, 7, 8, 6 | -1.8509 (9.27472) | 31.4853 (18.78336) | 49.3861 (14.33838) | 49.1721 (30.22147)
  Day 1, 6 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 6 hours, n=5, 7, 8, 6 | 3.3922 (6.75373) | 58.4446 (9.17750) | 70.8026 (8.26487) | 67.9378 (25.45192)
  Day 1, 8 hours, n=5, 7, 7, 6: number analyzed (Participants) | 5 | 7 | 7 | 6
  Day 1, 8 hours, n=5, 7, 7, 6 | 6.9714 (8.64363) | 58.4772 (9.97693) | 76.5366 (12.00112) | 69.8593 (23.77517)
  Day 1, 9 hours, n=1, 6, 0, 0: number analyzed (Participants) | 1 | 6 | 0 | 0
  Day 1, 9 hours, n=1, 6, 0, 0 | 18.8383 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 58.2218 (11.84589) |  |
  Day 1, 12 hours, n=4, 0, 7, 6: number analyzed (Participants) | 4 | 0 | 7 | 6
  Day 1, 12 hours, n=4, 0, 7, 6 | 1.1168 (9.94441) |  | 72.0336 (10.97106) | 72.4138 (28.39518)
  Day 1, 16 hours, n=4, 6, 8, 6: number analyzed (Participants) | 4 | 6 | 8 | 6
  Day 1, 16 hours, n=4, 6, 8, 6 | -1.9654 (4.50998) | 47.1603 (7.15517) | 79.1078 (8.03676) | 75.8997 (24.65609)
  Day 2, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 2, n=5, 7, 8, 6 | 5.8586 (11.64080) | 38.9846 (10.09414) | 67.5197 (8.13498) | 71.3820 (20.92599)
  Day 3, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 3, n=5, 7, 8, 6 | 8.4017 (21.57257) | 47.8814 (8.46678) | 77.5903 (8.78800) | 88.1872 (3.79283)
  Day 4, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 4, n=5, 7, 8, 6 | -2.2685 (9.15020) | 48.5169 (11.02802) | 82.0325 (10.26798) | 91.6139 (1.52341)
  Day 5, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 5, n=5, 7, 8, 6 | 9.4816 (10.25461) | 64.5703 (8.16040) | 88.1950 (6.33948) | 94.2542 (1.59484)
  Day 6, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, n=5, 7, 8, 6 | 4.6145 (5.61446) | 70.6624 (7.58163) | 89.9853 (4.21710) | 95.1333 (1.79263)
  Day 6, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, 1 hour, n=5, 7, 8, 6 | 8.0058 (7.53027) | 93.5215 (2.42406) | 91.9917 (2.78804) | 95.3978 (1.70448)
  Day 14, n=5, 6, 8, 4: number analyzed (Participants) | 5 | 6 | 8 | 4
  Day 14, n=5, 6, 8, 4 | 16.0448 (15.71866) | 18.3627 (15.59835) | 17.6415 (27.54591) | 38.7962 (17.92367)

17. Secondary Outcome: Relative Change From Baseline in Percentage (%) in CD8+ Cells
Description: Whole blood samples were collected and analyzed by flow cytometry. Day1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Relative change from baseline (%) was calculated as change from Baseline relative to Baseline in %. NA indicates that standard deviation could not be calculated for a single participant.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Percentage
  Day 1, 30 minutes, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 30 minutes, n=5, 7, 8, 6 | 1.4489 (5.86548) | 13.6045 (6.84553) | 18.4972 (10.57226) | 35.6721 (7.81791)
  Day 1, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 1 hour, n=5, 7, 8, 6 | 3.9227 (3.52082) | 23.2571 (8.77440) | 29.9262 (9.11960) | 37.1052 (15.47566)
  Day 1, 2 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 2 hours, n=5, 7, 8, 6 | 5.7591 (7.62243) | 29.7916 (10.08248) | 36.7030 (11.18167) | 48.2854 (10.33624)
  Day 1, 4 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 4 hours, n=5, 7, 8, 6 | 2.4574 (5.34591) | 27.9312 (15.06025) | 40.2754 (12.70208) | 41.5574 (26.91586)
  Day 1, 6 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 6 hours, n=5, 7, 8, 6 | 5.2570 (5.13603) | 50.6248 (8.12251) | 63.2777 (9.16749) | 61.0355 (22.44049)
  Day 1, 8 hours, n=5, 7, 7, 6: number analyzed (Participants) | 5 | 7 | 7 | 6
  Day 1, 8 hours, n=5, 7, 7, 6 | 3.0516 (5.05296) | 50.0586 (13.15793) | 64.0559 (8.96743) | 64.6389 (23.37406)
  Day 1, 9 hours, n=1, 6, 0, 0: number analyzed (Participants) | 1 | 6 | 0 | 0
  Day 1, 9 hours, n=1, 6, 0, 0 | 12.0124 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 47.3877 (10.18779) |  |
  Day 1, 12 hours, n=4, 0, 7, 6: number analyzed (Participants) | 4 | 0 | 7 | 6
  Day 1, 12 hours, n=4, 0, 7, 6 | 4.6297 (1.55778) |  | 63.0325 (11.60295) | 68.2523 (25.41788)
  Day 1, 16 hours, n=4, 6, 8, 6: number analyzed (Participants) | 4 | 6 | 8 | 6
  Day 1, 16 hours, n=4, 6, 8, 6 | 2.4031 (9.29601) | 36.5804 (11.00323) | 73.7619 (9.27676) | 73.7870 (23.65616)
  Day 2, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 2, n=5, 7, 8, 6 | 11.5153 (12.44266) | 32.3389 (17.53306) | 63.2076 (11.90764) | 68.8582 (23.13445)
  Day 3, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 3, n=5, 7, 8, 6 | 9.6580 (17.96579) | 38.6763 (10.50068) | 73.4518 (13.11370) | 86.3391 (4.07679)
  Day 4, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 4, n=5, 7, 8, 6 | 1.4965 (9.56563) | 39.4735 (13.72429) | 78.2797 (13.97813) | 89.7661 (2.38427)
  Day 5, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 5, n=5, 7, 8, 6 | 13.1690 (10.31403) | 55.7138 (7.92647) | 84.6850 (10.08105) | 92.6561 (1.66146)
  Day 6, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, n=5, 7, 8, 6 | 9.5352 (4.64977) | 62.6915 (6.12617) | 87.5358 (6.72558) | 93.6820 (1.51640)
  Day 6, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, 1 hour, n=5, 7, 8, 6 | 9.6315 (7.30255) | 90.8426 (2.43623) | 91.3298 (3.00883) | 93.9939 (1.50147)
  Day 14, n=5, 6, 8, 4: number analyzed (Participants) | 5 | 6 | 8 | 4
  Day 14, n=5, 6, 8, 4 | 21.2448 (18.40147) | 19.6382 (18.17904) | 20.1594 (27.60057) | 33.4359 (23.03254)

18. Secondary Outcome: Change From Baseline in Free CD3 on CD8+ Cells
Description: Whole blood samples were drawn and analyzed by flow cytometry. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. NA indicates that standard deviation could not be calculated for a single participant.
Time Frame: as for outcome 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Copies per cell
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Copies per cell
  Day 1, 30 minutes, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 30 minutes, n=5, 7, 8, 6 | -1570.2 (7996.97) | -17344.6 (8219.24) | -33177.1 (26046.74) | -46590.5 (14242.51)
  Day 1, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 1 hour, n=5, 7, 8, 6 | -5367.8 (4454.93) | -30170.0 (11702.96) | -52164.3 (25780.68) | -45971.2 (17371.50)
  Day 1, 2 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 2 hours, n=5, 7, 8, 6 | -7599.6 (9683.28) | -38063.3 (12268.28) | -64195.5 (30475.25) | -63303.5 (19743.02)
  Day 1, 4 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 4 hours, n=5, 7, 8, 6 | -2668.2 (7081.48) | -37523.3 (21827.29) | -70708.9 (35060.26) | -50216.3 (33433.24)
  Day 1, 6 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 6 hours, n=5, 7, 8, 6 | -7434.0 (6566.98) | -65821.7 (14778.18) | -109702.0 (36004.22) | -75299.7 (24515.25)
  Day 1, 8 hours, n=5, 7, 7, 6: number analyzed (Participants) | 5 | 7 | 7 | 6
  Day 1, 8 hours, n=5, 7, 7, 6 | -5118.8 (9260.84) | -64346.1 (16499.07) | -113884.9 (36548.70) | -79778.2 (25001.56)
  Day 1, 9 hours, n=1, 6, 0, 0: number analyzed (Participants) | 1 | 6 | 0 | 0
  Day 1, 9 hours, n=1, 6, 0, 0 | -14630.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | -62113.7 (17114.28) |  |
  Day 1, 12 hours, n=4, 0, 7, 6: number analyzed (Participants) | 4 | 0 | 7 | 6
  Day 1, 12 hours, n=4, 0, 7, 6 | -7671.0 (3453.02) |  | -111484.0 (37822.49) | -84085.8 (27533.48)
  Day 1, 16 hours, n=4, 6, 8, 6: number analyzed (Participants) | 4 | 6 | 8 | 6
  Day 1, 16 hours, n=4, 6, 8, 6 | -2398.0 (12735.14) | -48607.8 (17774.03) | -126378.6 (34284.38) | -91537.5 (23378.53)
  Day 2, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 2, n=5, 7, 8, 6 | -16282.6 (18931.53) | -42379.1 (25223.07) | -108857.0 (36292.51) | -85611.5 (24571.30)
  Day 3, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 3, n=5, 7, 8, 6 | -12613.4 (23082.56) | -50757.1 (16662.32) | -126037.9 (39171.31) | -112220.0 (20740.64)
  Day 4, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 4, n=5, 7, 8, 6 | -2479.6 (14120.73) | -52064.6 (22177.41) | -133794.1 (38684.37) | -116816.5 (22469.30)
  Day 5, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 5, n=5, 7, 8, 6 | -19504.4 (14161.40) | -72058.3 (13158.75) | -144613.4 (35791.57) | -120512.7 (22578.38)
  Day 6, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, n=5, 7, 8, 6 | -13905.4 (6365.89) | -81326.7 (14410.25) | -149202.1 (32099.88) | -121836.0 (22706.98)
  Day 6, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, 1 hour, n=5, 7, 8, 6 | -14414.4 (10131.25) | -118000.6 (18946.75) | -155565.6 (29776.06) | -122237.2 (22786.52)
  Day 14, n=5, 6, 8, 4: number analyzed (Participants) | 5 | 6 | 8 | 4
  Day 14, n=5, 6, 8, 4 | -30658.2 (25814.70) | -25656.7 (23202.59) | -34478.6 (46509.48) | -49846.8 (42800.88)

19. Secondary Outcome: Change From Baseline in Free CD3 on CD4+ Cells
Description: as for outcome 18
Time Frame: as for outcome 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Copies per cell
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Copies per cell
  Day 1, 30 minutes, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 30 minutes, n=5, 7, 8, 6 | 5529.0 (13037.93) | -26310.0 (15691.77) | -46612.6 (31524.47) | -61053.8 (16266.15)
  Day 1, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 1 hour, n=5, 7, 8, 6 | 2819.2 (8108.55) | -41955.9 (16287.89) | -68726.5 (33738.60) | -63524.8 (26817.94)
  Day 1, 2 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 2 hours, n=5, 7, 8, 6 | -5833.0 (17972.31) | -54111.1 (23197.46) | -86880.5 (37961.85) | -87013.2 (20852.00)
  Day 1, 4 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 4 hours, n=5, 7, 8, 6 | 2651.6 (14138.56) | -54076.3 (34638.82) | -101829.5 (45896.19) | -73042.7 (45129.43)
  Day 1, 6 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 6 hours, n=5, 7, 8, 6 | -5072.0 (11737.82) | -97871.0 (18824.51) | -143635.8 (41952.00) | -104097.7 (36063.45)
  Day 1, 8 hours, n=5, 7, 7, 6: number analyzed (Participants) | 5 | 7 | 7 | 6
  Day 1, 8 hours, n=5, 7, 7, 6 | -10668.4 (11325.47) | -97642.4 (17931.01) | -156878.1 (38450.32) | -107788.0 (34304.89)
  Day 1, 9 hours, n=1, 6, 0, 0: number analyzed (Participants) | 1 | 6 | 0 | 0
  Day 1, 9 hours, n=1, 6, 0, 0 | -31435.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | -98963.5 (25253.18) |  |
  Day 1, 12 hours, n=4, 0, 7, 6: number analyzed (Participants) | 4 | 0 | 7 | 6
  Day 1, 12 hours, n=4, 0, 7, 6 | -4958.5 (15637.79) |  | -150231.0 (46611.02) | -111627.8 (43965.70)
  Day 1, 16 hours, n=4, 6, 8, 6: number analyzed (Participants) | 4 | 6 | 8 | 6
  Day 1, 16 hours, n=4, 6, 8, 6 | 4546.3 (7628.46) | -79792.2 (16063.80) | -159376.9 (40492.21) | -117485.2 (35848.96)
  Day 2, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 2, n=5, 7, 8, 6 | -9071.4 (22730.36) | -64674.3 (14881.25) | -136989.0 (40208.17) | -111246.8 (30955.42)
  Day 3, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 3, n=5, 7, 8, 6 | -9750.2 (28173.66) | -80703.6 (19670.68) | -156782.3 (42746.51) | -141892.0 (28600.19)
  Day 4, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 4, n=5, 7, 8, 6 | 4442.8 (16258.54) | -81174.3 (21094.09) | -165042.3 (42878.04) | -147344.5 (28442.20)
  Day 5, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 5, n=5, 7, 8, 6 | -14696.4 (15969.14) | -107817.7 (16112.46) | -177310.9 (40876.20) | -151768.5 (30266.62)
  Day 6, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, n=5, 7, 8, 6 | -7848.0 (10416.76) | -118246.4 (17896.58) | -180424.5 (37325.84) | -153238.7 (30828.00)
  Day 6, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, 1 hour, n=5, 7, 8, 6 | -12708.6 (8424.98) | -156241.0 (14748.58) | -184362.0 (36070.44) | -153638.3 (30779.71)
  Day 14, n=5, 6, 8, 4: number analyzed (Participants) | 5 | 6 | 8 | 4
  Day 14, n=5, 6, 8, 4 | -25564.4 (24902.78) | -31243.3 (25714.52) | -37536.4 (55570.83) | -70890.5 (40581.96)

20. Secondary Outcome: Change From Baseline in Bound CD3 Copies on CD4+ Cells
Description: as for outcome 18
Time Frame: as for outcome 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Copies per cell
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Copies per cell
  Day 1, 30 minutes, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 30 minutes, n=5, 7, 8, 6 | -54.0 (103.13) | 29059.1 (15150.15) | 27538.5 (12441.29) | 28035.7 (14672.79)
  Day 1, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 1 hour, n=5, 7, 8, 6 | -10.2 (82.62) | 39472.3 (16401.81) | 43911.8 (14701.05) | 38406.5 (19297.11)
  Day 1, 2 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 2 hours, n=5, 7, 8, 6 | 27.6 (133.59) | 54116.3 (14159.80) | 56840.6 (15756.66) | 47028.2 (24507.94)
  Day 1, 4 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 4 hours, n=5, 7, 8, 6 | -50.4 (113.62) | 62635.7 (24380.73) | 54693.1 (16678.89) | 42730.2 (24609.04)
  Day 1, 6 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 6 hours, n=5, 7, 8, 6 | -77.4 (168.73) | 86518.1 (23953.89) | 74664.6 (5837.58) | 49078.8 (27502.89)
  Day 1, 8 hours, n=5, 7, 7, 6: number analyzed (Participants) | 5 | 7 | 7 | 6
  Day 1, 8 hours, n=5, 7, 7, 6 | 13.6 (203.64) | 86801.1 (24642.24) | 60435.0 (24147.90) | 51092.2 (25386.18)
  Day 1, 9 hours, n=1, 6, 0, 0: number analyzed (Participants) | 1 | 6 | 0 | 0
  Day 1, 9 hours, n=1, 6, 0, 0 | -36.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 55085.3 (14474.39) |  |
  Day 1, 12 hours, n=4, 0, 7, 6: number analyzed (Participants) | 4 | 0 | 7 | 6
  Day 1, 12 hours, n=4, 0, 7, 6 | -2.8 (188.70) |  | 57280.0 (7920.20) | 34176.7 (22339.84)
  Day 1, 16 hours, n=4, 6, 8, 6: number analyzed (Participants) | 4 | 6 | 8 | 6
  Day 1, 16 hours, n=4, 6, 8, 6 | 62.3 (278.48) | 33286.2 (10303.10) | 46080.4 (7254.50) | 28515.0 (13537.67)
  Day 2, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 2, n=5, 7, 8, 6 | -120.8 (157.70) | 14676.3 (4819.20) | 27994.6 (7683.11) | 23777.3 (10220.98)
  Day 3, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 3, n=5, 7, 8, 6 | -56.4 (209.56) | 15982.6 (5415.43) | 23383.9 (7380.09) | 19095.8 (4142.74)
  Day 4, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 4, n=5, 7, 8, 6 | -199.0 (221.61) | 12522.1 (4472.75) | 17241.8 (3135.36) | 14843.3 (3645.33)
  Day 5, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 5, n=5, 7, 8, 6 | -31.4 (334.36) | 9679.6 (3432.37) | 5748.1 (2499.44) | 6979.3 (4026.59)
  Day 6, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, n=5, 7, 8, 6 | -103.4 (138.02) | 4856.7 (4683.55) | 3671.9 (1663.91) | 4700.3 (2723.61)
  Day 6, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, 1 hour, n=5, 7, 8, 6 | -22.2 (385.45) | 15972.9 (4968.41) | 4262.9 (2221.09) | 4658.3 (2789.87)
  Day 14, n=5, 6, 8, 4: number analyzed (Participants) | 5 | 6 | 8 | 4
  Day 14, n=5, 6, 8, 4 | -111.2 (227.74) | -874.7 (2068.49) | 688.0 (513.77) | 1506.3 (2330.70)

21. Secondary Outcome: Change From Baseline in Bound CD3 Copies on CD8+ Cells
Description: as for outcome 18
Time Frame: as for outcome 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Copies per cell
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Copies per cell
  Day 1, 30 minutes, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 30 minutes, n=5, 7, 8, 6 | 10.8 (168.01) | 20952.1 (9089.08) | 22141.3 (9619.64) | 23518.7 (12011.07)
  Day 1, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 1 hour, n=5, 7, 8, 6 | 85.8 (253.77) | 28365.3 (9711.56) | 34147.9 (11206.05) | 32445.0 (16424.62)
  Day 1, 2 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 2 hours, n=5, 7, 8, 6 | 101.2 (265.29) | 35963.7 (6942.11) | 42469.1 (13977.93) | 38510.7 (19273.02)
  Day 1, 4 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 4 hours, n=5, 7, 8, 6 | 76.0 (209.69) | 41046.0 (14859.06) | 43492.8 (15811.41) | 43477.2 (28963.40)
  Day 1, 6 hours, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 1, 6 hours, n=5, 7, 8, 6 | -130.8 (273.14) | 68337.3 (22986.71) | 77279.4 (14115.24) | 55195.8 (27523.26)
  Day 1, 8 hours, n=5, 7, 7, 6: number analyzed (Participants) | 5 | 7 | 7 | 6
  Day 1, 8 hours, n=5, 7, 7, 6 | -60.4 (242.85) | 68342.4 (27742.23) | 70935.4 (10888.79) | 50511.3 (25067.72)
  Day 1, 9 hours, n=1, 6, 0, 0: number analyzed (Participants) | 1 | 6 | 0 | 0
  Day 1, 9 hours, n=1, 6, 0, 0 | 50.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 46941.7 (15418.31) |  |
  Day 1, 12 hours, n=4, 0, 7, 6: number analyzed (Participants) | 4 | 0 | 7 | 6
  Day 1, 12 hours, n=4, 0, 7, 6 | -9.8 (267.43) |  | 56618.7 (8092.43) | 40765.8 (21505.21)
  Day 1, 16 hours, n=4, 6, 8, 6: number analyzed (Participants) | 4 | 6 | 8 | 6
  Day 1, 16 hours, n=4, 6, 8, 6 | 30.8 (353.27) | 35124.7 (31051.56) | 47713.4 (7841.92) | 29753.0 (15501.29)
  Day 2, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 2, n=5, 7, 8, 6 | -41.2 (263.98) | 14020.9 (2453.61) | 26096.8 (5228.98) | 22559.8 (13107.67)
  Day 3, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 3, n=5, 7, 8, 6 | -29.0 (351.20) | 13502.1 (6856.86) | 19841.5 (4986.13) | 20615.5 (11473.73)
  Day 4, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 4, n=5, 7, 8, 6 | -90.0 (332.42) | 11065.7 (5053.88) | 17923.5 (2476.65) | 17694.8 (8442.57)
  Day 5, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 5, n=5, 7, 8, 6 | 49.0 (412.48) | 7781.6 (2908.32) | 7139.3 (2922.96) | 9209.5 (5670.67)
  Day 6, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, n=5, 7, 8, 6 | -59.4 (291.67) | 4706.7 (4049.36) | 4795.4 (2544.14) | 6093.3 (3673.79)
  Day 6, 1 hour, n=5, 7, 8, 6: number analyzed (Participants) | 5 | 7 | 8 | 6
  Day 6, 1 hour, n=5, 7, 8, 6 | 10.0 (566.43) | 20140.3 (6799.16) | 6011.8 (3638.55) | 6167.5 (3965.76)
  Day 14, n=5, 6, 8, 4: number analyzed (Participants) | 5 | 6 | 8 | 4
  Day 14, n=5, 6, 8, 4 | -84.4 (321.06) | -783.3 (1407.22) | 564.3 (374.97) | 1082.3 (1638.04)

22. Secondary Outcome: Number of Participants With Anti-drug Antibody Binding
Description: Samples were analyzed for the presence of anti-Otelixizumab antibodies using a validated immunoelectrochemiluminescent (ECL) assay.
Time Frame: Day-1, Month 3 and Month 6
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
Number analyzed (Participants) | 5 | 9 | 8 | 7
Participants
  Day -1, Negative | 3 | 9 | 8 | 6
  Day-1, Positive | 2 | 0 | 0 | 1
  Month 3, Negative | 3 | 0 | 0 | 0
  Month 3, Positive | 2 | 9 | 8 | 7
  Month 3, Newly Positive | 0 | 9 | 8 | 6
  Month 3, Negative who were Positive previously | 0 | 0 | 0 | 0
  Month 6, Negative | 3 | 0 | 0 | 0
  Month 6, Positive | 2 | 8 | 8 | 7
  Month 6, Newly Positive | 0 | 0 | 0 | 0
  Month 6, Negative who were Positive previously | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: On treatment serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment up to 36 months.
Description: Safety population was used. Safety population comprised of all participants who received at least one dose of a study treatment.
Arm/Group | Placebo | Otelixizumab 9 mg | Otelixizumab 18 mg | Otelixizumab 27 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/5 | 2/9 | 1/8 | 1/7
Other Adverse Events (participants affected / at risk) | 5/5 | 9/9 | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | Otelixizumab 9 mg (N=9) | Otelixizumab 18 mg (N=8) | Otelixizumab 27 mg (N=7)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | Otelixizumab 9 mg (N=9) | Otelixizumab 18 mg (N=8) | Otelixizumab 27 mg (N=7)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (434) | 9 (646) | 8 (210) | 7 (622)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (118) | 9 (380) | 7 (360) | 7 (215)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (25) | 9 (45) | 8 (25) | 7 (32)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 3 (3)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (7) | 8 (16) | 7 (15)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (9) | 6 (10) | 7 (12)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (7) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 3 (4) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0) | 2 (2) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (6) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival recession (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (12) | 7 (14) | 7 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (5) | 6 (10) | 4 (7) | 5 (11)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (4) | 3 (4) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 5 (5) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 3 (3) | 5 (5) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 4 (8) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 6 (11) | 4 (8)
Fatigue (General disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Chills (General disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Application site scab (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram QT Prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Repetitive strain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (6) | 2 (2) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 1 (1) | 3 (6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT02000817/SAP_000.pdf
  • Study Protocol (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT02000817/Prot_001.pdf